CLINICAL TRIAL: NCT06885424
Title: A Long-Term Follow-Up Study of Participants Treated With A2 Biotherapeutics (A2Bio) Gene Therapy (GT) Products
Brief Title: A Long-Term Follow-Up Study of Participants Treated With A2 Biotherapeutics (A2 Bio) Gene Therapy (GT) Products
Acronym: DESCENT-1
Status: Enrolling by invitation | Type: Observational
Sponsor: A2 Biotherapeutics Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: A2B101-201
Record Dates: First submitted 2025-03-12; First posted 2025-03-20 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Solid Tumor Cancer; Solid Tumor, Unspecified, Adult; Colorectal Carcinoma; Colorectal Carcinoma (CRC); Non Small Cell Lung Cancer; Small Cell Lung Cancer ( SCLC ); Pancreatic Cancer; NSCLC; Mesothelioma; Ovarian Cancer; Ovarian Carcinoma; Head and Neck (HNSCC); Head and Neck Cancer; Renal Cell Carcinoma (Kidney Cancer); Triple Negative Breast Cancer (TNBC)
Keywords: CAR T Cell Therapy; Gene Therapy
MeSH Terms: conditions — Colorectal Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Pancreatic Neoplasms; Mesothelioma; Ovarian Neoplasms; Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms; Carcinoma, Renal Cell; Kidney Neoplasms; Triple Negative Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood and Peripheral Blood Mononuclear Cells (PBMCs) will be analyzed for biomarkers and safety testing if required. No further genetic testing will be performed on these samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants that received A2 Bio GT products
  Interventions: Other: No additional intervention administered in this long term follow-up study

INTERVENTIONS:
Other: No additional intervention administered in this long term follow-up study — Safety follow-up for A2 Bio GT products administered in a previous interventional study

SUMMARY:
This protocol is to ensure consistent long-term follow-up for delayed safety events in participants who received A2 Bio gene therapy (GT) products.

DETAILED DESCRIPTION:
This is a long-term follow-up study designed to evaluate delayed safety events and long-term efficacy of A2 Bio GT products for participants who received any amount of A2 Bio GT products in a previous interventional study. No further interventional treatment is administered in this study.

Participants will enroll in this long-term follow-up study upon completion of 2 years of follow-up in the assigned interventional study in which they received treatment. Participants will be followed for up to 15 years after administration of A2 Bio GT product. This study will collect long-term safety and efficacy data as outlined by the FDA guidance for long-term follow-up for GT products.

ELIGIBILITY:
Inclusion Criteria:

1. Received any amount of A2 Bio GT product on a previous A2 Bio interventional study
2. Able to provide written informed consent for this long-term follow-up study
3. Able to comply with study requirements

Exclusion Criteria:

1. There are no specific exclusion criteria for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants previously treated on a A2 Bio GT study
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-08-31 (Estimated); Primary Completion 2030-03-31 (Estimated); Study Completion 2040-03-31 (Estimated)

PRIMARY OUTCOMES:
Long-term safety of previous A2 Bio GT treatment | 15 years post treatment with A2 Bio GT product
  Long-term safety of previous A2 Bio GT treatment as determined by incidence of adverse events (AEs)

SECONDARY OUTCOMES:
Overall survival | 15 years post treatment with A2 Bio GT product
  The time from dosing of A2 Bio GT product to the date of death from any cause
Long-term durability of clinical effect of previous A2 Bio GT treatment | 15 years post treatment with A2 Bio GT product
  Long-term durability of clinical effect of previous A2 Bio GT treatment as measured by duration of response (DOR)
Progression Free Survival (PFS) | 15 years post treatment with A2 Bio GT product
  Time from dosing of A2 Bio GT products to the date of disease progression or death from any cause, whichever occurs earlier
Incidence of RCL detected in blood | 15 years post treatment with A2 Bio GT product
  RCL will be tested on blood by ddPCR as applicable based on FDA guidance

OTHER OUTCOMES:
Progression Free Survival 2 (PFS2) | 15 years post treatment with A2 Bio GT product
  Time from start of the next line of treatment after A2 Bio product to the date of disease progression or death from any cause, whichever occurs earlier
Persistence of of A2 Bio GT | 5 years post treatment with A2 Bio GT product
  Amount of A2 Bio GT present in patients treated with A2 Bio GT as assessed by Polymerase Chain Reaction (PCR) (or similar method) on participant blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Eric Ng, MD, Study Director — A2 Biotherapeutics
Locations (2):
- United States (2):
  - Mayo Clinic, Rochester, Minnesota
  - NYU Langone Medical Center, New York, New York

REFERENCES:
- See also: A2 Bio Website — http://www.a2bio.com